CLINICAL TRIAL: NCT00048464
Title: A Phase I/II Study of Xcellerated T Cells After Autologous Peripheral Blood Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: T Cell Immunotherapy for Multiple Myeloma Patients Undergoing a Bone Marrow Transplant
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xcyte Therapies (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT003
Record Dates: First submitted 2002-10-31; First posted 2002-11-04 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2005-03

CONDITIONS: Multiple Myeloma
Keywords: Immunotherapy; T Cell Therapy; Peripheral Blood Stem Cell Transplant; Bone marrow transplant; Adoptive immunotherapy; Xcellerate
MeSH Terms: conditions — Multiple Myeloma

INTERVENTIONS:
Procedure: Infusion of Activated & Expanded Autologous T Cells

SUMMARY:
Patients will have immune cells collected and then expanded outside of the body. Patients will undergo standard treatment with high dose chemotherapy followed by peripheral blood stem cell transplantation. Three days following the transplant, patients will receive an infusion of a large number of expanded immune cells. The goal of the study will be to determine the safety as well as potential efficacy of this treatment.

DETAILED DESCRIPTION:
This Phase I/II clinical study is designed to examine the safety of Xcellerated T Cells, an activated, autologous T cell product, in study subjects undergoing an autologous peripheral blood stem cell transplant for the treatment of multiple myeloma. Thirty-five patients will be treated. Patients must have undergone induction therapy prior to study registration, and may not have progressed following induction therapy or any other prior therapy for myeloma.

Patients will undergo a steady state leukapheresis (Xcellerate Leukapheresis) to obtain peripheral blood mononuclear cells that will be used to produce Xcellerated T Cells. During the Xcellerate Process, T cells will be activated and expanded ex vivo by co-stimulation with anti-CD3 and anti-CD28 monoclonal antibodies covalently attached to super-paramagnetic microbeads. While the Xcellerated T Cells are being produced at Xcyte Therapies, patients will be treated with a standard mobilization regimen consisting of cyclophosphamide and filgrastim (Neupogen; G-CSF), followed by a second leukapheresis for collection of peripheral blood stem cells. Patients will be treated with a standard high-dose chemotherapy regimen for multiple myeloma consisting of single agent melphalan (200mg/m2). Patients will then receive their peripheral blood stem cells followed by post-transplant filgrastim for neutrophil recovery. Three days (Day 3) following stem cell infusion, patients will receive a single dose Xcellerated T Cells.

ELIGIBILITY:
Patient Inclusion Criteria

* Previous diagnosis of multiple myeloma based on standard criteria. Tests need not be performed within 30 days of registration.
* Durie-Salmon Stage II or III disease at any time since diagnosis
* Induction therapy with a minimum of 3 cycles of chemotherapy or 3 months of high-dose corticosteroids without progressive disease. (Note: no glucocorticoids are allowed within 3 weeks of registration; see exclusion criteria.)
* Measurable serum and/or urine M-protein from prior to induction therapy documented and available
* Lymphocyte subsets by flow cytometry demonstrating CD3+ >= 10% of the peripheral white blood cell count, and CD4+/CD8+ >= 0.30. Test must be obtained following completion of induction therapy.
* Meets all institutional criteria for and has institutional approval to undergo autologous peripheral blood stem cell transplantation
* Age >= 18 years old and <=70 years old
* ECOG performance status of 0 or 1
* Life expectancy > 6 months
* Females of child-bearing potential must have a negative serum bHCG test and be willing to use effective contraception (i.e. a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) up to Day 180.
* Negative test results for current/active infection with HIV-1, HIV-2, hepatitis B, and hepatitis C within 60 days of registration.(Antibody, antigen and nucleic acid tests acceptable, depending on institutional standards.)
* Corrected serum calcium < 11 mg/dL, and no evidence of symptomatic hypercalcemia. (Corrected serum calcium is calculated by adding 0.8 mg/dL to the measured serum calcium for every 1 g/dL that the serum albumin falls below 4.0 g/dL.)
* Serum total bilirubin and SGPT (ALT) < 2.0 times the upper limit of normal
* Serum creatinine < 2.0 mg/dL
* No detectable human anti-mouse antibody (HAMA) titer, and no history of allergies to mice or murine (mouse) proteins
* The patient must be able to comprehend and have signed the informed consent

Patient Exclusion Criteria

* Diagnosis of any of the following cancers:
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein] and skin changes)
* Non-secretory myeloma
* Plasma cell leukemia
* Diagnosis of amyloidosis
* Progression or relapse presently or in the past, during or following therapy for multiple myeloma
* Previous hematopoietic stem cell transplantation
* Use of corticosteroids (glucocorticoids) within 21 days of registration
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents within seven days of registration
* Participation in any clinical trial, within four weeks prior to registration on this trial, which involved an investigational drug or device
* History of malignancy other than multiple myeloma within five years of registration, except adequately treated basal or squamous cell skin cancer. Any other exceptions must be discussed with Xcyte Therapies' Medical Monitor prior to registration.
* History of an autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosis) requiring systemic treatment. Hypothyroidism without evidence of Grave's Disease or Hashimoto's thyroiditis is permitted.
* Evidence of spinal cord compression
* Major organ system dysfunction including (but not limited to): New York Heart Association Class III or IV, pulmonary disease requiring the use of inhaled steroids or bronchodilators, renal, hepatic, gastrointestinal, neurologic, or psychiatric dysfunction which would impair patient's ability to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2002-10

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Hackensack University, Hackensack, New Jersey

REFERENCES:
- [Background] Levine BL, Bernstein WB, Aronson NE, Schlienger K, Cotte J, Perfetto S, Humphries MJ, Ratto-Kim S, Birx DL, Steffens C, Landay A, Carroll RG, June CH. Adoptive transfer of costimulated CD4+ T cells induces expansion of peripheral T cells and decreased CCR5 expression in HIV infection. Nat Med. 2002 Jan;8(1):47-53. doi: 10.1038/nm0102-47. PMID 11786906
- [Background] Thomas AK, June CH. The promise of T-lymphocyte immunotherapy for the treatment of malignant disease. Cancer J. 2001 Nov-Dec;7 Suppl 2:S67-75. PMID 11777267
- [Background] June CH. Can't get any help? New approaches for adoptive immunotherapy of cancer. J Immunother. 2001 Sep-Oct;24(5):389-91. No abstract available. PMID 11696694
- [Background] Frohlich, M., Grosmaire, L., Xu, J., Rasmussen, A., Roehrs, H., Lindgren, R., Ferrand, C., Tiberghien, P., Leis, J., and Bonyhadi, ML: Xcellerate: a novel autologous T cell immunotherapeutic approach for the treatment of B-cell chronic lymphocytic leukemia (B-CLL). The IX International Workshop on CLL.2002.
- [Background] Li Q, Yu B, Grover AC, Zeng X, Chang AE. Therapeutic effects of tumor reactive CD4+ cells generated from tumor-primed lymph nodes using anti-CD3/anti-CD28 monoclonal antibodies. J Immunother. 2002 Jul-Aug;25(4):304-13. doi: 10.1097/00002371-200207000-00002. PMID 12142553